CLINICAL TRIAL: NCT07215325
Title: The Effects of Doxycycline on Inflammation and the Microbiome: 'Flipping the Script' on STI PEP
Brief Title: Got Doxy- 'Flipping the Script' on STI PEP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Colleen Kelley, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009355; 1R01AI192319-01 (NIH); 2025P009920 (Other: Emory IRB)
Record Dates: First submitted 2025-10-03; First posted 2025-10-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sexually Transmitted Infections (STI)
Keywords: Doxycycline post-exposure prophylaxis (doxy-PEP); Gut inflammation; Prevention; PEP; STI
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Doxycycline; Observation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxycycline 200mg (Experimental): Males with HIV infection on antiretroviral therapy or without HIV infection on HIV pre-exposure prophylaxis who are not taking doxy-PEP will be enrolled and randomized to take 12 weeks of doxycycline 200 mg by mouth three times weekly.
  Blood and rectal mucosal samples will be collected before the initiation of doxycycline.
  Interventions: Drug: Doxycycline monohydrate 200 mg
- Observation with biological sampling (Active Comparator): Males with HIV infection on antiretroviral therapy or without HIV infection on HIV pre-exposure prophylaxis who are not taking doxy-PEP will receive standard of care and will undergo biological sampling.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Doxycycline monohydrate 200 mg — Doxycycline monohydrate 200 mg (two 100 mg tablets) is used to treat or prevent infections that are strongly suspected to be caused by bacteria. Doxycycline monohydrate is an antimicrobial drug indicated for the treatment of bacterial infections, including sexually transmitted diseases. Centers for Disease Control and Prevention (CDC) recommends its use as post-exposure prophylaxis (PEP).
  Blood and rectal mucosal samples will be collected before doxycycline is initiated. Participants will be instructed to take 200 mg of doxycycline by mouth every Monday, Wednesday, and Friday. Additional doses of doxycycline will be permitted on other days if sex without a condom occurs per CDC guidance. After 12 weeks of at least three-weekly doxycycline, blood and rectal mucosal samples will be collected for immunologic and microbiome/resistome assays.
  Other Names: Doxycycline
  Arms: Doxycycline 200mg
Other: Observation — Standard of care. Blood and rectal mucosal samples.
  Other Names: Standard of Care
  Arms: Observation with biological sampling

SUMMARY:
This study is being done to test the effects of doxycycline on inflammation and the bacteria in the body in people with HIV and in people on HIV pre-exposure prophylaxis. This drug is approved by the Food and Drug Administration (FDA) for the treatment of bacterial infections.

The study team will investigate whether the drug has additional effects on inflammation or on the bacteria that live in the body.

DETAILED DESCRIPTION:
This project aims to determine the potential anti-inflammatory and microbiome effects of doxycycline when used as post-exposure prophylaxis (Doxy PEP) for sexually transmitted infections (STIs).

This study is important in the field of research because it allows the investigators to define the systemic and gut anti-inflammatory, microbiome, and resistome effects of doxycycline when used as post-exposure prophylaxis (Doxy PEP) for sexually transmitted infections. The study population that this study seeks to enroll consists of healthy people assigned male at birth, with and without HIV, who are willing to undergo study procedures.

Study procedures will include the collection of medical history, as well as biological specimen sampling, such as blood and rectal tissue biopsies.

The duration of this clinical trial for study participants will be approximately 12 weeks. This will include five in-person visits lasting about 45 minutes to 1 hour (including two biopsy visits).

This study will utilize data specimen banking for future research.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Assigned male sex at birth
* Good general health as assessed by a clinician at the screening study visit
* For people with HIV, on suppressive antiretroviral therapy for at least 6 months with the most recent viral load documented <50 copies/ml and the most recent cluster of differentiation 4 (CD4)>300cells/ul
* For people without HIV, taking oral daily, oral on-demand, or injectable pre-exposure prophylaxis for at least 3 months at the time of enrollment, with plans to continue for the duration of the study
* Additional criteria apply

Exclusion Criteria:

* Severe/uncontrolled comorbidities that could influence immune outcomes (e.g., diabetes, hypertension, co-infections), as assessed by the investigator.
* History of inflammatory bowel disease (IBD) or other inflammatory, infiltrative, infectious, or vascular condition involving the lower GI tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel.
* Known allergy to doxycycline
* Use of any antibiotics within 3 months before screening
* Significant lab abnormalities at baseline visit for rectal biopsies,
* Continued need for the following medications during the study:

  1. Aspirin
  2. Warfarin, heparin (LMW or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
  3. Any form of rectally administered agent besides products (lubricants or douching) used for sexual intercourse
  4. NSAIDS within 72 hours of rectal sampling procedures
* Continued need for, or use during the 90 days before enrollment, of the following medications:

  1. Systemic immunomodulatory agents
  2. Supraphysiologic doses of corticosteroids, except for short-course corticosteroids <7 days duration at the discretion of the investigator. (Gender affirming hormone therapy is not exclusionary.)
  3. Use of experimental medications, vaccines, or biologicals in the 12 months before enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Composite inflammation score | Baseline and 12 weeks after the start of doxycycline administration
  A composite inflammation score in the blood and rectal secretions before and after doxy-PEP will be calculated for each participant: +1 point for each proinflammatory cytokine (IP-10, IL-1β, tumor necrosis factor (TNF-α), Monocyte chemoattractant protein-1 (MCP-1), IL-17A, IL-6, interferon (IFN-γ), IL-12p70, IL-8) that was in the top quartile concentration and -1 point for each anti-inflammatory cytokine (IL-4, IL-10), T-cell growth factor (TGF-β1) that was in the top quartile concentration for a maximum score of 9 and minimum score of -3.

SECONDARY OUTCOMES:
Tetracycline (TCN) Gene Abundance | Baseline and 12 weeks after the start of doxycycline administration
  TCN gene-level abundance will be normalized using reads per kilobase per genome equivalent (RPKG), calculated from filtered contigs and estimated genome equivalents (MicrobeCensus). RPKG values will be summed by resistance class, sub-class (e.g., inactivation, target modification, efflux), and by host assignment (pathogen vs. commensal). Group differences in mean TCN RPKG values will be evaluated using non-parametric permutation tests.
Estimated mass of antimicrobial resistance (AMR) Genes | Baseline and 12 weeks after the start of doxycycline administration
  To benchmark normalized abundance, the mass of AMR genes will be estimated using spike-in controls (ZymoBIOMICS). This will provide a quantitative measure of the total AMR gene burden per sample. Group differences in total AMR gene mass will be tested using non-parametric permutation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System (non-CRN), Atlanta, Georgia
  - Hope Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published for this study will be made available for sharing after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: The research team will share de-identified participant data after publication of the primary results manuscript, anticipated on September 15, 2030. Data will be available indefinitely.
Access Criteria: Interested investigators may request de-identified data for secondary analyses and/or meta-analyses by contacting Dr. Kelley via email and completing a data use agreement (DUA) with Emory University.